CLINICAL TRIAL: NCT06320561
Title: Stroke-induced Muscular Changes and Their Relation to Clinical Impairments and Gait Recovery in the First 12 Weeks After Stroke.
Brief Title: Muscular Changes in the First 12 Weeks After Stroke.
Acronym: StrIMuC12
Status: Not yet recruiting | Type: Observational
Sponsor: Vrije Universiteit Brussel (Other)
Collaborators: University Ghent (Other); Research Foundation Flanders (Other)
Responsible Party: Principal Investigator, Eva Swinnen, Assistant professor, Vrije Universiteit Brussel
Other Study IDs: 23485_StrIMuC12
Record Dates: First submitted 2024-01-12; First posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Stroke
Keywords: Muscular changes; m. rectus femoris; m. gastrocnemius medials; Lower limb impairment; Gait recovery; Subacute phase; 3DfUS; sEMG; Dynamic ultrasound
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients in the first 3 months after stroke: Inclusion criteria:
  Adults (≥ 18 years old) Diagnosed with a first-ever stroke (as defined by WHO) Stroke onset ≤ 1 week (± 3 days) Able to provide written or verbal informed consent at admission Presence of gait problems as a consequence of the stroke (FAC≤4)
  Exclusion criteria:
  Presence of other neurological or orthopedic problems present prior to, or not caused as a direct consequence of, the stroke leading to impaired gait.
  Modified Ranking scale pre-stroke > 1/6, meaning presence of slight disability before the stroke.
  Presence of severe comorbidities (e.g. osteoporosis, cardiovascular instability or chronic obstructive pulmonary disease).
  Cerebellar or bilateral stroke. Presence of severe deficits in communication, memory or understanding precluding informed consent.
  Interventions: Other: Longitudinal prospective cohort study

INTERVENTIONS:
Other: Longitudinal prospective cohort study — Patients after stroke who meet the in- and exclusion criteria will be examined 4 times during the first 3 months after their stroke.

SUMMARY:
The investigators will use 3D freehand ultrasound to investigate changes in muscle morphology of the paretic m. rectus femoris and m. gastrocnemius medialis during the first 3 months after stroke. Additionally, 2D ultrasound and surface EMG will be synchronized to examine muscle activation and morphological changes resulting from this activation. Clinical tests will be conducted on the same test occasions to objectify lower limb impairment and gait recovery. As such, the investigators will explore the relationship between the muscle specific changes and functional recovery.

DETAILED DESCRIPTION:
During this longitudinal study, patients who suffer their first-ever stroke will be included within the first week after their stroke (if the inclusion criteria are met). Thereafter, each participant will be assessed at four pre-determined time-points: week 1, 5, 8 and 12 after stroke.

On each of the four time-points, the investigators will assess muscle specific parameters of the affected m. rectus femoris (RF) and m. gastrocnemius medialis (GM), together with clinical tests to assess lower limb impairment (Fugl-Meyer Assessment for the lower limb and the Tardieu scale) and gait parameters (10-meter walk test). Specifically, muscle specific parameters will be investigated using 3D freehand ultrasound (3DfUS) and combined dynamic 2D US and surface electromyography (sEMG). Such assessments will help us characterize the electromechanical properties of these muscles, their time-related trajectories and the relationship with the recovery of gait and lower limb function after stroke. At the end of the investigation period, after 3 months, patients who can walk independently will perform a 3D gait analysis. As such, the relationship between changes in muscle specific parameters and the eventual gait quality at the end of the investigation period will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥ 18 years old)
* Diagnosed with a first-ever stroke (as defined by WHO)
* Stroke onset ≤ 1 week (± 3 days)
* Able to provide written or verbal informed consent at admission
* Presence of gait problems as a consequence of the stroke (FAC≤4)

Exclusion Criteria:

* Presence of other neurological or orthopedic problems present prior to, or not caused as a direct consequence of, the stroke leading to impaired gait.
* Modified Ranking scale pre-stroke > 1/6, meaning presence of slight disability before the stroke.
* Presence of severe comorbidities (e.g. osteoporosis, cardiovascular instability or chronic obstructive pulmonary disease).
* Cerebellar or bilateral stroke.
* Presence of severe deficits in communication, memory or understanding precluding informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Persons who suffer their first-ever stroke (ischaemic or hemorrhagic) will be investigated during the subacute phase after the stroke (i.e. first 3 months).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Functional Ambulation Categories (FAC)-score | Frequency: week 1, 5, 8 and 12 after stroke
  Scores ranging from 0 (not able to walk) to 5 (independent ambulator who can walk freely on any surface)
Muscle volume | Frequency: week 1, 5, 8 and 12 after stroke
  Through 3D freehand ultrasound (3DfUS)
Cross-sectional area (CSA) | Frequency: week 1, 5, 8 and 12 after stroke
  Through 3D freehand ultrasound (3DfUS)
Physiological cross-sectional area (pCSA) | Frequency: week 1, 5, 8 and 12 after stroke
  Through 3D freehand ultrasound (3DfUS)
Muscle tickness | Frequency: week 1, 5, 8 and 12 after stroke
  Through 3D freehand ultrasound (3DfUS)
Fascicle length | Frequency: week 1, 5, 8 and 12 after stroke
  Through 3D freehand ultrasound (3DfUS)
Muscle length | Frequency: week 1, 5, 8 and 12 after stroke
  Through 3D freehand ultrasound (3DfUS)
Tendon length | Frequency: week 1, 5, 8 and 12 after stroke
  Through 3D freehand ultrasound (3DfUS)
Pennation angle | Frequency: week 1, 5, 8 and 12 after stroke
  Through 2D ultrasound
Echo Intensity | Frequency: week 1, 5, 8 and 12 after stroke
  Through 2D ultrasound
Dynamic muscle morphology | Frequency: week 1, 5, 8 and 12 after stroke
  Dynamic 2D ultrasound used to investigate the changes in cross-sectional area (CSA) en fascicle length
Change in cross-sectional area | Frequency: week 1, 5, 8 and 12 after stroke
  Through dynamic 2D ultrasound
Change in fascicle length | Frequency: week 1, 5, 8 and 12 after stroke
  Through dynamic 2D ultrasound
Average root mean square (RMS) | Frequency: week 1, 5, 8 and 12 after stroke
  Through surface electromyography (sEMG)
Peak root mean square (RMS) | Frequency: week 1, 5, 8 and 12 after stroke
  Through surface electromyography (sEMG)
Muscle strength | Frequency: week 1, 5, 8 and 12 after stroke
  Assessed with a handheld dynamometer (Nm)
Spasticity | Frequency: week 1, 5, 8 and 12 after stroke.
  Assessed with the Tardieu Scale. Scores ranging from 0 (no resistance throughout passive movement) to 5 (immobile joint).
Lower limb motor impairment | Frequency: week 1, 5, 8 and 12 after stroke.
  Fugl-Meyer Assessment of the lower limb (FMA LL). Scores ranging from 0 to 34 (no impairment present).
Spatiotemporal gait parameters | Frequency: week 1, 5, 8 and 12 after stroke.
  Patients will perform the 10-meter walk test while wearing the GaitUp sensors.
Gait quality | Frequency: only at week 12.
  Gait profile score (index number in degrees (°)), calculated from the lower limbs' kinematics (3D gait analysis). A higher score means more deviation of the expected (normal) gait pattern.

SECONDARY OUTCOMES:
TWIST-score | Within first week after stroke
  TWIST gait prediction model scores will be calculated to externally validate this model.
Knee extension strength | Frequency: only during the first assessment (week 1).
  Medical Research Council knee extension. Scores ranging from 0 (no muscular activity) to 5 (normal strength).
Balance | Frequency: only during the first assessment (week 1)
  Berg Balance Scale. Scores ranging from 0 (Severe balance deficits) to 56 (normal balance).

CONTACTS AND LOCATIONS:
Overall Officials: Eva Swinnen, Professor, Principal Investigator — Vrije Universiteit Brussel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Smith MC, Barber AP, Scrivener BJ, Stinear CM. The TWIST Tool Predicts When Patients Will Recover Independent Walking After Stroke: An Observational Study. Neurorehabil Neural Repair. 2022 Jul;36(7):461-471. doi: 10.1177/15459683221085287. Epub 2022 May 18. PMID 35586876